CLINICAL TRIAL: NCT06525766
Title: Single Arm Pilot Trial of Adaptive Therapy (AT) With Capecitabine for the Treatment of Metastatic Estrogen Receptor Positive, Hormone Refractory Breast Cancer
Brief Title: Adaptive Therapy With Capecitabine for Treatment of Metastatic ER Positive, HER2 Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC230303; NCI-2024-06184 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-009851 (Other: Mayo Clinic Institutional Review Board); MC230303 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Estrogen-receptor-positive Breast Cancer; Metastatic HER2-Negative Breast Carcinoma; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling; Capecitabine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (capecitabine) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Drug: Capecitabine; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial evaluates the effect of capecitabine on tumor response using imaging and tumor markers to adjust dose (adaptive therapy) in patients with estrogen receptor (ER) positive, HER2 negative breast cancer that has spread from where it first started to other areas in the body (metastatic). Capecitabine is in a class of medications called antimetabolites. It is taken up by tumor cells and breaks down into fluorouracil, a substance that kills tumor cells. Adaptive therapy with capecitabine based on tumor burden response may slow or stop the growth of tumor cells in patients with metastatic ER positive, HER2 negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the feasibility of adaptive therapy (AT) in hormone receptor positive metastatic breast cancer, defined as the number of patients who can achieve AT modification for 2 or more cycles.

SECONDARY OBJECTIVES:

I. To evaluate time to progression in patients receiving capecitabine AT defined as the interval between treatment start and tumor progression, or death in patients with no evidence of disease progression.

II. Assess overall survival in patients receiving capecitabine as adaptive therapy.

III. Evaluate patient related outcomes by measuring quality of life and global health status of patients on AT using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core 30 questionnaire EORTC QLQ C-30.

IV. Evaluate adverse events secondary to capecitabine using Common Terminology Criteria for Adverse Events (CTCAE) grading system version 5.0.

V. Assess feasibility and accuracy of radiologic 3 dimensional (3D) volumetric approach in measuring target lesions.

EXPLORATORY OBJECTIVES:

I. Assess circulating tumor deoxyribonucleic acid (DNA) (ctDNA) as a low-cost alternative to imaging for measuring tumor burden.

II. Identify gene signatures that could predict response and identify mechanisms of resistance to capecitabine using next generation sequencing technology, including:

IIa. Whole exome DNA sequencing from ctDNA at baseline (day 0) and end of treatment; IIb. Whole transcriptome ribonucleic acid (RNA) sequencing from ctDNA at and at baseline (day 0) and end of treatment.

III. ctDNA quantification is optional at day 1 (D-1).

OUTLINE:

INITIAL STANDARD PHASE: Patients receive standard dose of capecitabine orally (PO) twice daily (BID) on days 1-14 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients whose disease has responded or remains stable after 2 cycles continue to the Adaptive Phase.

ADAPTIVE PHASE: Patients receive 50% reduced dose of capecitabine PO BID on days 1-14 of each cycle. Patients undergo blood sample collection every cycle and computed tomography (CT) every other cycle for disease response assessment. Patients whose disease burden decreases < 10% on CT or blood begins receiving an additional 50% reduced dose of capecitabine PO BID on days 1-14 of each cycle. Patients whose disease burden is stable on CT or blood continue receiving initial Adaptive Phase dose of capecitabine PO BID on days 1-14 of each cycle. Patients whose disease burden increases > 10% on CT or blood begin receiving a 50% dose increase in capecitabine PO BID on days 1-14 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo blood sample collection, CT or magnetic resonance imaging (MRI), and bone scan if indicated on study.

After completion of study treatment, patients are followed up every 3 months for up to 3 years from time of registration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histological confirmation of estrogen-receptor positive (ER+), HER2-negative overexpression or amplification negative as per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines, metastatic breast cancer
* Measurable disease. Bone only disease allowed if associated with soft tissue component that is measurable by Response Evaluation Criteria is Solid Tumors (RECIST) 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Hemoglobin ≥ 9.0 g/dL (obtained ≤ 14 days prior to registration), no transfusions allowed ≤ 14 days prior to registration
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 14 days prior to registration)
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 14 days prior to registration)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained ≤ 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (≤ 5 x ULN for patients with liver involvement) (obtained ≤ 14 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy (obtained ≤ 14 days prior to registration)
* Calculated creatinine clearance ≥ 45 ml/min using the Cockcroft-Gault formula (obtained ≤ 14 days prior to registration)
* Negative serum or urine pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential only. NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to provide mandatory blood specimens for correlative research
* Ability to undergo re-staging CT scans as required by the protocol
* Willing to return to enrolling institution at the specified frequency for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Prior chemotherapy or use of antibody drug conjugate in the metastatic setting
* Any of the following, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Any of the following prior therapies:

  * Major surgery ≤ 3 weeks prior to registration
  * Radiation therapy ≤ 2 weeks prior to registration
* Evidence of visceral crisis or impending cord compression
* Evidence of uncontrolled brain metastasis requiring whole brain irradiation or intervention
* Uncontrolled intercurrent illness including, but not limited to:

  * ongoing or active infection
  * symptomatic congestive heart failure
  * unstable angina pectoris
  * uncontrolled cardiac arrhythmia
  * chronic oxygen dependence
  * respiratory failure
  * or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy ≤ 3 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
* If there is a history of prior malignancy, they must not be receiving other cancer specific treatment. Except for antiestrogen treatment (aromatase inhibitors or selective estrogen modulators) for their cancer are permitted if they meet other eligibility criteria. Denosumab and zoledronic acid, are permitted as established adjunct therapies per guidelines
* History of myocardial infarction ≤ 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Patients known to have certain homozygous or compound heterozygous dihydropyrimidine dehydrogenase (DPYD) variants that result in complete absence of deoxypyridinoline (DPD) activity
* History of severe hypersensitivity reactions to fluorouracil or capecitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-10-15 (Estimated); Study Completion 2030-10-15 (Estimated)

PRIMARY OUTCOMES:
Ability to achieve adaptive therapy (AT) | Up to 5 years
  Will be assessed by the proportion of patients (%) who are able to receive 2 or more cycles of AT with capecitabine divided by the total number of patients who have entered the AT phase of treatment (have stable or responsive disease).

SECONDARY OUTCOMES:
Time to progression | At registration to disease progression up to 5 years
  Time to progression will be defined as the time from registration to the earliest date of documentation of disease progression.
Overall survival (OS) | At registration to death up to 5 years
  OS will be defined as the time from registration to death due to any cause.
Cumulative dose | Up to 5 years
  The cumulative dose of capecitabine administered per patient will be assessed across patients receiving AT.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study drug
  The maximum grade for each type of AE will be recorded for each patient. Adverse events will be categorized according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Quality of life - EORTC-QLQ-C30 | Up to 5 years
  Will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30), a 30-question survey that measures the quality of life of cancer patients. The questionnaire has a score range of 0 to 100 points, with, higher scores indicating a better level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Lida A. Mina, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials